CLINICAL TRIAL: NCT03026283
Title: The Value of Fractional Flow Reserve Derived From Coronary CTA and in the Triage of Low to Intermediate Risk Chest Pain Patients: Design: Single Center Prospective Clinical Trial; Target Disease: Coronary Artery Disease
Brief Title: The Value of CT Fractional Flow Reserve
Acronym: VFFRCTA
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-765-LHH
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Angina, Stable Chest Pain
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 1: HeartFlow CT-FFR Arm: All patients who consent will receive HeartFlow CT-FFR and medically acceptable care based on the study protocol, commonly accepted standards of care, and the patients condition.
  Interventions: Device: HeartFLow CT-FFR

INTERVENTIONS:
Device: HeartFLow CT-FFR — Patients receiving CCTA to diagnose stable chest pain or stable angina will receive CT-FFR to estimate rate of flow through the coronary arteries. The rate of flow will be compared to the rate found on Invasive FFR (the gold standard) if the subject receives invasive FFR.
  Other Names: Noninvasive CT-FFR, FFR-CT, Noninvasive FFR-CT

SUMMARY:
Coronary Computed Tomography Angiogram (CCTA) is a non-invasive imaging modality that has high sensitivity and negative predictive value for the detection of coronary artery disease (CAD). The main limitations of CCTA are its poor specificity and positive predictive value, as well as its inherent lack of physiologically relevant data on hemodynamic significance of coronary stenosis, a data that is provided either by non-invasive stress tests such as myocardial perfusion imaging (MPI) or invasively by measurement of the Fractional Flow Reserve (FFR). Recent advances in computational fluid dynamic techniques applied to standard CCTA are now emerging as powerful tools for virtual measurement of FFR from CCTA imaging (CT-FFR). These techniques correlate well with invasively measured FFR [1-4]. The primary purpose of this study is to evaluate the incremental benefit CT-FFR as compared to CCTA in triaging chest pain patients in outpatient settings who are found to have obstructive CAD upon CCTA (> 30% and < 90% stenosis). Invasive FFR and short term clinical outcomes (90 days) will be correlated with each diagnostic modality in order to evaluate positive and negative predictive value of each when used incrementally with CCTA.

This will be an observational trial in which patients will undergo a CCTA, as part of routine care. If the patient consents to participate in the study and is found to have coronary stenosis of 30% to 90%, based on the cardiologist's reading, the CCTA study will be sent to HeartFlow, a vendor that will provide a computerized FFR reading, based on the CCTA study. If the noninvasive FFR diagnosis indicates obstructive disease, the patient will be recommended to undergo cardiac catheterization with invasive FFR.

As CCTA utilization increases, the need to train additional imaging specialists will increase. This study will assess the capability of FFR-CT to enhance performance on both negative and positive predictive value for less experienced readers by providing feedback based on CT-FFR evaluation. CCTA readers will be grouped in two categories: those with more than 10 years reading experience and those with less than 10 years reading experience. Each CCTA will be read by a less experienced and a more experienced reader. Results from each reader will be correlated with each other and with the CT-FFR and invasive FFR results.

DETAILED DESCRIPTION:
CCTA is increasingly becoming a preferred non-invasive imaging modality because of its high sensitivity and negative predictive value for the detection of CAD. It has been shown to be a robust imaging modality for evaluation of chest pain, and is associated with decreased unnecessary hospital admission, length of stay, major adverse cardiovascular event rates, recidivism rates, and downstream resource utilization compared to standard evaluation [5]. While findings so far are highly suggestive of CCTA's significance as a gatekeeper for Invasive Coronary Angiography (ICA) by ruling out obstructive CAD, fewer than half of obstructive stenosis identified by CCTA are ischemia-causing, signifying its poor positive predictive value and inherent lack of physiological information [6-8]. Consequently, utilization of CCTA has not entirely averted need for downstream testing for functional assessment of CCTA-detected obstructive lesions either by stress testing or ICA. Recently a major treatment modality, associated with the use of CCTA, has become available that offers promise for improving positive predictive value and physiological relevant hemodynamic data. Advances in computational fluid dynamic techniques applied to standard CCTA are now emerging as a powerful tool for virtual measurement of FFR from CCTA imaging (CT-FFR). This techniques correlate well with invasively measured FFR [1-4]. CT-FFR is not an investigational agent, having been approved by FDA in November, 2014. However, more work is necessary to delineate the patient population that could derive maximal benefit from this new technology.

While few publications regarding the use of CT-FFR specifically address the cost of diagnostic work-up for obstructive disease, it is clear that the cost structure resulting from changes in diagnostic testing will also change. Deferral or avoidance of cardiac catheterization and nuclear stress testing will likely yield significant reductions in the cost of the diagnostic testing.

From 1/1/2009 to 3/31/2015 our team introduced and operated a CCTA Chest Pain triage program for low to intermediate risk patients at Stony Brook University Hospital ED and non-emergency outpatient services, the only tertiary care hospital in Suffolk County. Concurrently, we established a registry to monitor patient outcomes for all patients receiving CCTA at Stony Brook Medicine. Our registry contained nearly 15,000 patient CCTA procedures. Our major registry study established the effectiveness of CCTA as an imaging modality for evaluating Emergency Department chest pain in a cost efficient manner with a false negative rate less than 1% [5]. However, our registry reflects the poorer positive predictive values documented by other industry studies [6-8].

False positive workup results in the necessity of performing cardiac catheterization on patients at risk for obstructive disease based on assessment with current standard of care (combined screening with CCTA and stress MPI). Reduction in the rate of false positive testing would lead to reduction in risk from invasive procedures and radiation exposure to patients and reduced cost to the health care system.

Several medical institutions currently use HeartFlow CT-FFR as standard of care for evaluating obstructive disease. Generally, the standard of care at these institutions is to refer patients who are 30 to 90 percent obstructed by CCTA and who have reduction of flow <= to 0.8 that is deemed to be medical significant by the attending cardiologist to Invasive FFR. HeartFlow has reported to us confidentially that this routine use of CT-FFR has resulted in a 54% reduction in false positive rate as compared to use of CCTA alone.

The purpose of this study is to evaluate the incremental benefit of Fractional Flow Reserve derived from CCTA (FFR-CT) compared invasive FFR as the gold standard for patients with obstructive disease (> 30% and < 90% stenosis). This study will also assess the capability of CT-FFR to enhance performance on both negative and positive predictive value for less experienced readers by providing feedback based on CT-FFR evaluation.

This will be a prospective observational clinical trial designed to evaluate the incremental benefit of virtual FFR measured from CCTA, compared to invasive FFR and CCTA for the detection of flow-limiting coronary stenosis, as defined by invasive FFR <0.8 and vessel diameter of >=2mm.

572 consecutive patients who present to Lenox Hill Hospital Outpatient Clinics for CCTA due to chest pain or stable angina over a ten month period and meeting the study inclusion criteria are eligible for the study (Figure 1). Our team will employ CCTA-appropriateness criteria to ensure proper selection of patients, derived from the Appropriate Use Criteria for Cardiac Computed Tomography published in 2010 and jointly authored by multiple societies including American College of Cardiology Foundation (ACCF), Society for Cardiovascular Computed Tomography (SCCT), and American College of Radiology (ACR) [10]. FFR-CT measurements will be performed by a core laboratory in a blinded fashion. All eligible patients will undergo 64-slice or greater multi detector CCTA and CT-FFR measurements. The severity of the stenosis will be determined on site by level III CCTA readers. Patients with obstructive lesions of (30% to 90% stenosis) will be referred for Stress-MPI, per SOC protocol, and CT-FFR. Patients with positive Stress-Myocardial Perfusion Imaging (MPI) and CCTA (50% - 70%%) or positive CCTA (71% to 90%) will be referred for undergo ICA with invasive FFR measurement in accordance to accepted guidelines and established practice standard. They will also received CT-FFR. Those patients with invasively measured FFR<0.8 and with vessel diameter of >= 2mm, or those who require revascularizations based on invasively estimated stenosis severity will be considered to have flow-limiting obstructive CAD, while the rest will be considered to have non-flow limiting obstructive CAD (if also >50% stenosis on ICA). If stenosis severity turns out to be < 50% after ICA (the gold standard), we will conclude that these patients have non-obstructive CAD. (Figure 1). Patients with 30% to 49% obstructive disease, according to CCTA, will be referred to optimal follow up care only. Any in this group who have positive CT-FFR will return for ICA with invasive FFR measurement, and follow the protocol for those with 50% to 90% obstruction.

Defining an event as performance of ICA when no intervention is necessary, we expect to compare event rates for patients treated with CCTA and FFR-CT, using t-tests and a multivariate, risk adjusted 90 day hazard model with 95% confidence interval. Our null hypothesis is that outcomes will not vary regardless of which testing is used to assess obstructive disease. Our alternative hypothesis is that evaluation with FFR-CT as oppose to CTTA will change the event rate. We will also correlate noninvasive and invasive FFR studies.

We will assess inter-observer reliability of the two reader cohorts' (> 10 years experience and less than 10 years experience) readings for CCTA and CT-FFR.. We will also assess the nondiagnostic rate for CT-FFR exams as compared to independent quality ratings of CCTA scans by the scan reader. Scans will be rated as excellent, good, adequate, or non-diagnostic. Non-diagnostic exams will not be sent to CT-FFR. For those sent to CT-FFR we will compare the percentage of non-diagnostic exams to the percentage of non-diagnostic for CT-FFR, and we will also correlate exam results by level of obstruction.

ELIGIBILITY:
1. Inclusion Criteria:
2. Capable of giving informed consent.
3. Able to cooperate with the technician performing the procedure.
4. Patient must have Body Mass Index (BMI) <= 50.
5. Patients must have non-ST Elevation Myocardial Infarction (STEMI) Electrocardiogram (EKG) without acute changes.
6. Patients must present to Research Institution with medically necessary appointment for CCTA for the purpose of evaluation of coronary stenosis for the provisional diagnoses of chest pain or angina or angina equivalent.
7. Patients must be able to take nitroglycerin and beta blockers. -
8. Patients must be 18 years of age or older.

Exclusion Criteria:

1. Patients must not have a history of coronary stenting or coronary artery bypass graft.
2. Patients must not have severe or end stage renal disease as diagnosed as estimated glomerular filtration rate (eGFR)<50.
3. Patients must not have a BMI>50.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We reviewed a patient registry of 7,001 Stony Brook Medicine CCTA from 2011 to 2014,(work from our team members' prior research). About one third of the subjects were stable chest pain patients.
Sampling Method: Non-Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Poon, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koo BK, Erglis A, Doh JH, Daniels DV, Jegere S, Kim HS, Dunning A, DeFrance T, Lansky A, Leipsic J, Min JK. Diagnosis of ischemia-causing coronary stenoses by noninvasive fractional flow reserve computed from coronary computed tomographic angiograms. Results from the prospective multicenter DISCOVER-FLOW (Diagnosis of Ischemia-Causing Stenoses Obtained Via Noninvasive Fractional Flow Reserve) study. J Am Coll Cardiol. 2011 Nov 1;58(19):1989-97. doi: 10.1016/j.jacc.2011.06.066. PMID 22032711
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266
- [Background] Liu HY, Chen JR, Hung HC, Hsiao SY, Huang ST, Chen HS. Urinary fluoride concentration in children with disabilities following long-term fluoride tablet ingestion. Res Dev Disabil. 2011 Nov-Dec;32(6):2441-8. doi: 10.1016/j.ridd.2011.07.016. Epub 2011 Aug 5. PMID 21820860
- [Background] Niska R, Bhuiya F, Xu J. National Hospital Ambulatory Medical Care Survey: 2007 emergency department summary. Natl Health Stat Report. 2010 Aug 6;(26):1-31. PMID 20726217
- [Background] Poon M, Cortegiano M, Abramowicz AJ, Hines M, Singer AJ, Henry MC, Viccellio P, Hellinger JC, Ferraro S, Poon A, Raff GL, Voros S, Farkouh ME, Noack P. Associations between routine coronary computed tomographic angiography and reduced unnecessary hospital admissions, length of stay, recidivism rates, and invasive coronary angiography in the emergency department triage of chest pain. J Am Coll Cardiol. 2013 Aug 6;62(6):543-52. doi: 10.1016/j.jacc.2013.04.040. Epub 2013 May 15. PMID 23684682
- [Background] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693
- [Background] Meijboom WB, Meijs MF, Schuijf JD, Cramer MJ, Mollet NR, van Mieghem CA, Nieman K, van Werkhoven JM, Pundziute G, Weustink AC, de Vos AM, Pugliese F, Rensing B, Jukema JW, Bax JJ, Prokop M, Doevendans PA, Hunink MG, Krestin GP, de Feyter PJ. Diagnostic accuracy of 64-slice computed tomography coronary angiography: a prospective, multicenter, multivendor study. J Am Coll Cardiol. 2008 Dec 16;52(25):2135-44. doi: 10.1016/j.jacc.2008.08.058. PMID 19095130
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Taylor AJ, Cerqueira M, Hodgson JM, Mark D, Min J, O'Gara P, Rubin GD; American College of Cardiology Foundation Appropriate Use Criteria Task Force; Society of Cardiovascular Computed Tomography; American College of Radiology; American Heart Association; American Society of Echocardiography; American Society of Nuclear Cardiology; North American Society for Cardiovascular Imaging; Society for Cardiovascular Angiography and Interventions; Society for Cardiovascular Magnetic Resonance; Kramer CM, Berman D, Brown A, Chaudhry FA, Cury RC, Desai MY, Einstein AJ, Gomes AS, Harrington R, Hoffmann U, Khare R, Lesser J, McGann C, Rosenberg A, Schwartz R, Shelton M, Smetana GW, Smith SC Jr. ACCF/SCCT/ACR/AHA/ASE/ASNC/NASCI/SCAI/SCMR 2010 appropriate use criteria for cardiac computed tomography. A report of the American College of Cardiology Foundation Appropriate Use Criteria Task Force, the Society of Cardiovascular Computed Tomography, the American College of Radiology, the American Heart Association, the American Society of Echocardiography, the American Society of Nuclear Cardiology, the North American Society for Cardiovascular Imaging, the Society for Cardiovascular Angiography and Interventions, and the Society for Cardiovascular Magnetic Resonance. J Am Coll Cardiol. 2010 Nov 23;56(22):1864-94. doi: 10.1016/j.jacc.2010.07.005. PMID 21087721
- See also: NIH National heart, Lung and Blood Institute, What are the risks of cardiac catheterization — https://www.nhlbi.nih.gov/health-topics/cardiac-catheterization

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 1/24/2017 to 6/13/2018 patients seen in the Cardiology ambulatory care service for CCTA to be evaluated for the diagnosis of obstructive disease, and who were evaluated as low to intermediate risk for obstructive disease, and who were symptomatic were offered the opportunity to participate in the study.
Pre-assignment Details: To participate, patients were required to complete the CCTA, and on exam have no Cardiac stenting or bypasses as determined by medical history provided by the patient and review of CCTA scan.
Groups:
- Initial CCTA: All patients who consent will receive CCTA and medically acceptable care based on commonly accepted standards of care, and the patient's condition. The results of the CCTA will determine whether the patient receives FFR-CT or optimal medical care.
- Optimal Medical Care After CCTA: Patients who receive a CCTA and for whom the results are normal or less than 30% obstructive disease, will be recommended for optimal medical care. This care is the commonly accepted standard of care as recommended by the patient's referring physician. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- FFR-CT After CCTA: Patients for whom CCTA results show 30% of more obstructive disease will be referred for FFR-CT. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- Optimal Medical Care After FFR-CT: Patients with negative FFR-CT and CCTA results showing 30 to 49% obstructive disease will be recommended for optimal medical care with their Cardiologist, and patients with positive FFR-CT and CCTA results showing 30 to 49% obstructive disease will be recommended for stress testing. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- Stress Testing After FFR-CT: Patients with 50% to 69% obstructive disease on CCTA and negative FFR-CT will be recommended for stress testing. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- ICA/Diagnostic Catheterization After FFR-CT: Patients with 50 to 69% obstructive disease and positive FFR-CT will be referred for diagnostic catheterization and patients with 70% obstructive disease or greater by CCTA will be referred for diagnostic catheterization. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- Optimal Care After Stress Test: Patients who undergo stress testing will be referred to optimal medical care if the results are negative. (The referring physician will make all treatment decisions, and may not follow the recommendation provided by the study team).
- ICA/Diagnostic Catheterization After Stress Test: Patients who undergo stress testing will be referred to diagnostic catheterization if the result is positive.
Period: CCTA Diagnosis
Arm/Group | Initial CCTA | Optimal Medical Care After CCTA | FFR-CT After CCTA | Optimal Medical Care After FFR-CT | Stress Testing After FFR-CT | ICA/Diagnostic Catheterization After FFR-CT | Optimal Care After Stress Test | ICA/Diagnostic Catheterization After Stress Test
Started | 586 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 572 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — CCTA not performed as planned | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Optimal Medical Care/FFR-CT Diagnosis
Arm/Group | Initial CCTA | Optimal Medical Care After CCTA | FFR-CT After CCTA | Optimal Medical Care After FFR-CT | Stress Testing After FFR-CT | ICA/Diagnostic Catheterization After FFR-CT | Optimal Care After Stress Test | ICA/Diagnostic Catheterization After Stress Test
Started (Note: Number of participants to start period is not equal to number who completed previous period.) | 0 | 289 | 280 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 286 | 265 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 15 | 0 | 0 | 0 | 0 | 0
Not completed — Screen Failure: Enrollment Criteria | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — FFRCT Nondiagnostic | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0
Period: Optimal Care/Stress Test/ICA
Arm/Group | Initial CCTA | Optimal Medical Care After CCTA | FFR-CT After CCTA | Optimal Medical Care After FFR-CT | Stress Testing After FFR-CT | ICA/Diagnostic Catheterization After FFR-CT | Optimal Care After Stress Test | ICA/Diagnostic Catheterization After Stress Test
Started (Participants diagnosed to receive optimal care, or recommended for stress test diagnosis or ICA) | 0 | 0 | 0 | 128 | 52 | 101 | 0 | 0
Completed (Participants who followed recommendation provided after consultation with referring physician.) | 0 | 0 | 0 | 108 | 14 | 73 | 0 | 0
Not Completed | 0 | 0 | 0 | 20 | 38 | 28 | 0 | 0
Not completed — Referring MD ordered diagnostic cath | 0 | 0 | 0 | 8 | 11 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9 | 2 | 2 | 0 | 0
Not completed — Referring MD ordered stress test | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Referring MD used only optimal med care | 0 | 0 | 0 | 0 | 25 | 19 | 0 | 0
Period: Optimal Care/ICA Diagnostic Cath
Arm/Group | Initial CCTA | Optimal Medical Care After CCTA | FFR-CT After CCTA | Optimal Medical Care After FFR-CT | Stress Testing After FFR-CT | ICA/Diagnostic Catheterization After FFR-CT | Optimal Care After Stress Test | ICA/Diagnostic Catheterization After Stress Test
Started (Participants recommended for ICA or optimal medical care after stress testing) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The initial enrollment number was 586. However, 14 patients did not receive CCTA, and three additional patients became screen failures, due to medical conditions revealed on the CCTA screen. Therefore the total reported is 569.
Arm/Group | 1: HeartFlow CT-FFR Arm
Number analyzed (Participants) | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289
  Male | 280
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72
  Not Hispanic or Latino | 497
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 79
  White | 295
  More than one race | 136
  Unknown or Not Reported | 0
Indication [Count of Participants; unit: Participants]
  Angina (Typical) | 62
  Angina (Atypical) | 284
  Noncardiac Chest Pain | 1
  Dyspnea | 170
  Angina Status Unknown | 2
  Angina Status None | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg per meters squared] — Participants height and weight were recorded upon enrollment and BMI was calculated. Population: Height and weight data was not recorded on enrollment for one participant.
  kg per meters squared
    number analyzed (Participants) | 568
    (all) | 28.23 (6.15)
Diabetes [Count of Participants; unit: Participants] — Participants who reported having diabetes Population: Three study participants did not respond when asked if they were diabetic.
  Participants
    number analyzed (Participants) | 566
    (all) | 117
Hypertension [Count of Participants; unit: Participants] — Participants were asked upon enrollment if they had been diagnosed with hypertension that required treatment. Population: Two participants were unable to report whether they had been diagnosed and were being treated for hypertension,
  Participants
    number analyzed (Participants) | 567
    (all) | 337
Hyperlipidemia [Count of Participants; unit: Participants] — Participants were asked upon enrollment whether they had be diagnosed with hyperipidemia requiring medical treatment. Population: Five study participants were unable to report upon enrollment whether they had been diagnosed with hyperlipidemia.
  Participants
    number analyzed (Participants) | 564
    (all) | 312
Smoking History [Count of Participants; unit: Participants] — Participants were asked if they were a current smoker, had smoke in the past but quit, or had never smoked. Population: 9 Participants did not disclosed their smoking history.
  Participants
    Never Smoked: number analyzed (Participants) | 560
    Never Smoked | 364
    Former Smoker: number analyzed (Participants) | 560
    Former Smoker | 157
    Current Smoker: number analyzed (Participants) | 560
    Current Smoker | 39

OUTCOME MEASURES:

1. Primary Outcome: Comparison of CCTA Alone to FFR-CT After CCTA
Description: To evaluate sensitivity, specificity, positive and negative predictive value for FFR-CT after CCTA vs. CCTA alone, using invasive FFR as the gold standard.
Time Frame: Up to 1 year from the study initiation will be required to enroll all study patients and obstain invasive and noninvasive FFR.
Population: All patients who received FFR-CT and Diagnostic Catheterization.
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- CCTA: .CCTA Alone
- FFR-CT After CCTA: FFR-CT After CCTA
Arm/Group | CCTA | FFR-CT After CCTA
Number analyzed (Participants) | 97 | 97
percent
  Sensitivity | 90.97 [79.70 to 96.62] | 92.73 [82.41 to 97.98]
  Specifcity | 22.86 [10.42 to 40.14] | 69.71 [46.49 to 80.25]
  Positive Predictive Value | 64.47 [52.66 to 75.12] | 80.95 [69.09 to 89.75]
  Negative Predictive Value | 60.67 [49.75 to 70.87] | 84.62 [65.13 to 95.64]
Statistical Analysis 1: Comparison: CCTA vs FFR-CT After CCTA; Reference test is positive (test of sensitivity); Test type: Other; p = 1.00, Chi-squared — In order to evaluate the significance of sensitivity and specificity findings, we implement McNemar's test comparing sensitivity and specificity for CCTA alone and FFR-CT, assuming conditional dependence
Statistical Analysis 2: Comparison: CCTA vs FFR-CT After CCTA; Reference test is Negative; Test type: Other; p < 0.0047, Chi-squared — In order to evaluate the significance of sensitivity and specificity findings, we implement Mcnemar's test comparing sensitive and pscificity for CCTA and FFR-CT assuming dependence; McNemar's chi-squared = 8.00

2. Secondary Outcome: Inter-observer Reliability: Assessment of All Cases
Description: To evaluate differences in performance of readers of CCTA and CT-FFR based on years of experience. CCTA results were documented by the official reader, all of whom had less than 9 years experience reading CCTA. Independently the exams were reviewed by a second reader with more than 10 years experience reading CCTA. Due to an operational error, for 5 of the 572 cases that received CCTA, the detailed data was removed from the server before the second read. Therefore these cases were excluded from this analysis.
Time Frame: Up to 1 year will be required to obtain all reader evaluations for the study in order to asses inter-observer reliability.
Population: All patients who received CCTA, for whom scans were available for clinical review and review by the study's expert reader.
Measure: Mean (Standard Error); unit: percent agreement
Units Other Than Participants: CCTA Scans
Groups:
- CCTA Reading: Less Experienced Reader Vs. More Experience: All CCTA results were read by readers with fewer than10 years experience and who spent at least one full time day per week reading CCTA and FFR-CT. These are the official results performed during the course of care. We tested agreement with expert reader with more than 10 years experience, who supervised the practice and did not routinely perform daily clinical reads.
  The arm initially had 572 subjects who completed CCTA exams. However, detailed scan results for 5 patients were inadvertently removed from the server before the second reader could review, and therefore, could not be included in the analysis.
Arm/Group | CCTA Reading: Less Experienced Reader Vs. More Experience
Number analyzed (Participants) | 567
Number analyzed (CCTA Scans) | 567
percent agreement | 67.72 (0.0247)

3. Secondary Outcome: Inter - Observer Reliability: Assessment of at Least Mild Disease (30% Stenosis or More)
Description: To evaluate differences in performance of readers of CCTA and CT-FFR based on years of experience when assessing cases on which the official reading identified at least mild disease. Mild disease is defined as cases with 30% or more stenosis documented on CCTA reading. CCTA cases that cannot be read are treated as severe.)
Time Frame: as for outcome 2
Population: The less experienced reader read 271 of the CCTA scan as having Mild disease -- 30% obstructive disease or more. We compared these reading to the expert reader's assessment for the same cases.
Measure: Mean (Standard Error); unit: percent agreement
Groups:
- Less Experienced Reader Vs. More Experience: CCTA and FFR-CT results read by readers with fewer than10 years experience and who spent at least one full time day per week reading CCTA and FFR-CT. These are the official results performed during the course of care. We tested agreement with expert reader with more than 10 years experience.
Arm/Group | Less Experienced Reader Vs. More Experience
Number analyzed (Participants) | 271
percent agreement | 35.79 (0.0262)

4. Secondary Outcome: Inter - Observer Reliability: Assessment of at Least Moderate Disease (50% Stenosis or More on CCTA)
Description: To evaluate differences in performance of readers of CCTA and CT-FFR based on years of experience when assessing cases on which the official reading is at least moderate (50% stenosis on CCTA. CCTA cases that cannot be read are treated as severe.
Time Frame: as for outcome 2
Population: The less experienced reader called moderate stenosis or higher (50% or more stenosis) on 159 cases.
Measure: Mean (Standard Error); unit: percent agreement
Arm/Group | Less Experienced Reader Vs. More Experience
Number analyzed (Participants) | 159
percent agreement | 40.88 (0.0385)

5. Secondary Outcome: Inter - Observer Reliability: Assessment of Severe Disease is Diagnosesed on Official Read (70% or Greater)
Description: To evaluate differences in performance of readers of CCTA and CT-FFR based on years of experience when assessing cases with suspected severe disease on the official reading. (CCTAs that cannot be read are treated as severe).
Time Frame: as for outcome 2
Population: The population of patients expected to have severe of more (70% obstructive disease or more) on CCTA by less experienced reader interpretation.
Measure: Mean (Standard Error); unit: percent agreement
Arm/Group | Less Experienced Reader Vs. More Experience
Number analyzed (Participants) | 83
percent agreement | 51.81 (0.0422)

6. Secondary Outcome: Return Visits
Description: To identify factors influencing return visits within 90 days for all patients enrolled who received CCTA. While we are not aware of any documented incremental risks for adding FFR-CT to the evaluation process of coronary artery disease, this safety measure was designed to identify and evaluate all unplanned return events to ensure that they were not related to FFR-CT or to flaws in study design or operations.
Time Frame: Up to 15 months will be required to collect 90 day follow up information on all study participants.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: This is a safety measure to assess urgent and emergency returns for services within 90 days of the initial encounter. Emergency returns for Acute Myocardial Infarction or urgent need for revascularization, were evaluated by the study safety committee to determine whether participation in the study had contributed to major adverse event.
Arm/Group | All Study Participants
Number analyzed (Participants) | 572
Participants
  Direct Admit from CCTA | 4
  Urgent/Unplanned return within 90 days | 11
  No Unplanned/Urgent returns in 90 days | 557

7. Secondary Outcome: Return Visits -- Reasons for Return
Description: To identify factors influencing return visits within 90 days. All patient's who returned to the ED within 90 days of their initial visit were contacted for follow up. All their medical records were reviewed.
Time Frame: Up to 15 months will be required to collect 90 day follow up information on all study participants.
Population: Overall 15/572 (2.6%) patients returned for emergent visits. All outcomes may be viewed as being consistent with the diagnoses provided with CCTA and FFR-CT.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initially Referred for Cardiac Cath: These patients were referred for diagnostic Cath, because their CCTA was positive and their FFR-CT was positive.
- Patients Initially Referred for Stress Tesintg: These patients had Moderate (50 to 69% stenoisis) finding on CCTA with Negative FFR-CT. They were referred to stress testing by protocol. One patient underwent a negative diagnostic cardiac cath. One patient was treated and released fro the ED for chest pain.
- Referred for Optimla Medical Care After CCTA: These patients were referred to optimal medical care after CCTA. They returned to the Emergency Department with Chest Pain and were discharged after evaluation and noninvasive treatment.
Arm/Group | Patients Initially Referred for Cardiac Cath | Patients Initially Referred for Stress Tesintg | Referred for Optimla Medical Care After CCTA
Number analyzed (Participants) | 11 | 2 | 2
Participants
  Severe Disease Received Intervention | 11 | 0 | 0
  Nonobstructive Disease Went to Cardiac Cath | 0 | 1 | 0
  Nonobstructive Disease Discharged from ED | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: 90 days from the imaging encounter.
Description: Serious adverse events were major cardiac events (Acute Myocardial Infarction, death or emergency cardiac intervention). Other adverse events unnecessary exposure to invasive testing or higher risk health care environment, such as return to ED or unexpected referrals to diagnostic cardiac cath.
Groups:
- Patients Referred for Cardiac Intervention: Patients for whom Cardiac Catheterization was recommended after protocol testing.
- Patients Referred for Stress Tesing: Patients for whom stress testing was recommended after FFR-CT
- Patients Referred for Optimal Medical Care: Patients for whom optimal medical care was recommended after protocol testing.
Arm/Group | Patients Referred for Cardiac Intervention | Patients Referred for Stress Tesing | Patients Referred for Optimal Medical Care
All-Cause Mortality (participants affected / at risk) | 2/101 | 0/73 | 0/398
Serious Adverse Events (participants affected / at risk) | 1/101 | 1/73 | 0/398
Other Adverse Events (participants affected / at risk) | 0/101 | 2/73 | 2/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Referred for Cardiac Intervention (N=101) | Patients Referred for Stress Tesing (N=73) | Patients Referred for Optimal Medical Care (N=398)
Percutaneous Coronary Intevention (Cardiac disorders) | 1 (1) | 1 (1) | NA — Patients diagnosed with acute disease recommended to follow up with their referring physicians had chest pain and sent to ED by physician's recommendation before treatment was completed on an ambulatory basis. Received PCI and discharged home.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Referred for Cardiac Intervention (N=101) | Patients Referred for Stress Tesing (N=73) | Patients Referred for Optimal Medical Care (N=398)
Diagnostic Catheterization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — A patient with findings of mild nonobstructive disease was recommended for optimal medical care. However, after consultation with referring physician has negative diagnostic catheterization. Classified as unnecessary risk exposure adverse event.
Return to ED for Chest Pain (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) — 3 patients experience chest pain and came to ED. Patients were discharged home after treatment. Classified as unnecessary risk exposure adverse event.

LIMITATIONS AND CAVEATS:
This is an observational trial. The study team made recommendations to referring physicians after diagnostic work-up with CCTA and FFR-CT we performed. However, it was up to the referring physician as to whether to follow them.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03026283/Prot_SAP_000.pdf